CLINICAL TRIAL: NCT06562816
Title: Comparing Trypsin-Chymotrypsin and Naproxen Sodium for Post-endodontic Treatment Pain: a Randomized Controlled Trial
Brief Title: Comparing Trypsin-Chymotrypsin and Naproxen Sodium for Post-endodontic Treatment Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hafsa Zaki, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3376
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Effect of Drug
Keywords: Trypsin-Chymotrypsin; Naproxen Sodium; Symptomatic Irreversible Pulpitis; Acute Irreversible Pulpitis; Post-endodontic treatment pain; Root canal treatment; Proteolytic Enzyme
MeSH Terms: interventions — chymotrypsin, trypsin drug combination; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trypsin-Chymotrypsin (Experimental): This group will receive sealed envelopes containing oral formulations of Trypsin:Chymotryspin in the ratio of 6:1 with an enzymatic activity of 100000 A.U./tablet (Tab. Chymoral Forte) three times a day, 30 minutes before meals for 24 hours.
  Interventions: Drug: Trypsin-Chymotrypsin
- Naproxen Sodium (Active Comparator): The active control group will receive oral formulation of Naproxen Sodium 550mg (Tab. Synflex) twice a day, after meals for 24 hours.
  Interventions: Drug: Naproxen Sodium 550mg

INTERVENTIONS:
Drug: Trypsin-Chymotrypsin — 100000 IU
  Other Names: Chymoral Forte
  Arms: Trypsin-Chymotrypsin
Drug: Naproxen Sodium 550mg — 550mg
  Other Names: Synflex 550mg
  Arms: Naproxen Sodium

SUMMARY:
This study aims to compare the pain reduction efficacy of Trypsin-Chymotrypsin and Naproxen sodium after root canal treatment in patients with symptomatic irreversible pulpitis. A lot of patients suffer greatly from post endodontic treatment pain and have a fear of dental treatments due to the pain. Patients refuse to go to the dentists and neglect oral hygiene care. That's why it is very important to find an effective drug regimen to reduce this post treatment pain. The null hypothesis is that there will be no difference between the efficacy and mean pain scores of Trypsin-chymotrypsin and Naproxen Sodium for post-endodontic treatment pain. Conducted as a triple-blinded, parallel, randomized controlled trial, 100 patients will be randomly assigned to receive either Trypsin-Chymotrypsin or Naproxen sodium following standard root canal therapy. Pain levels will be assessed using a numerical rating scale at 1, 6, 12, and 24 hours post-treatment to evaluate the effectiveness of these two pain management modalities.

DETAILED DESCRIPTION:
i. Background Prevention or management of pain, especially after root canal treatment, is of utmost importance to Endodontists. Non-steroidal anti-inflammatory drugs (NSAIDs) have been the most commonly used pain reduction modality in cases of irreversible pulpitis, but they do come with certain demerits. A lot of other alternatives have been researched as better alternatives for NSAIDs. Trypsin- Chymotrypsin has been proven to be an effective pain reducer after endodontic therapy.

ii. Objective The objective of this study is to compare the pain reduction efficacy of Trypsin- Chymotrypsin and Naproxen sodium after root canal treatment.

iii. Methodology In this triple-blinded, parallel, randomized controlled trial, a total of 100 patients will be included who are coming to the Operative Dentistry department for root canal treatment for any tooth. The patient must have a history of symptomatic irreversible pulpitis. The patients will be randomly allocated into two groups. One group (n = 50 will be the Trypsin- Chymotrypsin group, and the second group (n = 50) will be the Naproxen sodium group (active control group). The root canal treatment will be performed as usual. The first group will receive Trypsin- Chymotrypsin 1:100000 and the second group will receive Naproxen Sodium 550mg in sealed envelopes. The intensity of post-operative pain will be evaluated using a numerical rating scale at 1 hour, 6 hours, 12 hours, and 24 hour intervals.

iv. Sequence Generation: Computer generated randomization using appropriate software (random.org) to assign the participants to trypsin-chymotrypsin or naproxen sodium group, ensuring a complete random allocation to each treatment arm, decreasing a risk of bias and enhancing the internal validity of the study.

v. Blinding: The participants, researcher and outcome assessors will be blinded in this research (triple blinded).

vi. Allocation Concealment: The allocation concealment will be achieved by packaging medicines in tightly sealed, opaque envelopes by a different person not conducting research or assessing outcomes. This process ensured that researchers involved in participant enrollment could not predict or influence the treatment assignment, reducing the risk of selection bias.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female, healthy patients (ASA class 1).
* Patients between the age group of 18-45 years.
* Patients who are appointed for endodontic treatment.
* Maxillary or mandibular teeth diagnosed with symptomatic irreversible pulpitis based on delayed responses to vitality tests.

Exclusion Criteria:

* Patients who will require emergency dental treatment.
* Teeth with any form of peri-apical lesion will be excluded.
* Patient who have taken analgesics within 24 hours prior to the treatment.
* Patients with known hypersensitivity or allergy to any of the study medications.
* Patients with any systemic disease such as uncontrolled diabetes, gastric ulcers, bleeding disorders, or cardiovascular problems.
* Pregnant or lactating women and pediatric patients.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in post-endodontic treatment pain score using Numeric Rating Scale | 24 hours
  The Numeric Rating Scale (NRS-11) is an eleven-point scale that ranges from 0, indicating no pain, to 10, representing the most severe pain the patient has ever encountered.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hafsa Zaki, Principal Investigator — DUHS
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
There is some information that can be sensitive to some patients. Sharing this data can compromise their confidentiality and cause a breach of their privacy. Anonymous data can be shared upon request.

REFERENCES:
- [Background] Mehrvarzfar P, Abbott PV, Saghiri MA, Delvarani A, Asgar K, Lotfi M, Karamifar K, Kharazifard MJ, Khabazi H. Effects of three oral analgesics on postoperative pain following root canal preparation: a controlled clinical trial. Int Endod J. 2012 Jan;45(1):76-82. doi: 10.1111/j.1365-2591.2011.01950.x. Epub 2011 Sep 8. PMID 21902704
- [Background] Hashem AAR, Abd El Sattar AA, Abdel Rahman TY. The Effect of Trypsin-Chymotrypsin on Postoperative Pain after Single Visit Endodontic Treatment: A Randomized Controlled Trial. J Endod. 2023 Mar;49(3):240-247. doi: 10.1016/j.joen.2022.12.010. Epub 2022 Dec 24. PMID 36574828
- [Background] Cooper SA, Desjardins P, Brain P, Paredes-Diaz A, Troullos E, Centofanti R, An B. Longer analgesic effect with naproxen sodium than ibuprofen in post-surgical dental pain: a randomized, double-blind, placebo-controlled, single-dose trial. Curr Med Res Opin. 2019 Dec;35(12):2149-2158. doi: 10.1080/03007995.2019.1655257. Epub 2019 Aug 27. PMID 31402718
- [Background] Tampi MP, Pilcher L, Urquhart O, Kennedy E, O'Brien KK, Lockhart PB, Abt E, Aminoshariae A, Durkin MJ, Fouad AF, Gopal P, Hatten BW, Lang MS, Patton LL, Paumier T, Suda KJ, Cho H, Carrasco-Labra A. Antibiotics for the urgent management of symptomatic irreversible pulpitis, symptomatic apical periodontitis, and localized acute apical abscess: Systematic review and meta-analysis-a report of the American Dental Association. J Am Dent Assoc. 2019 Dec;150(12):e179-e216. doi: 10.1016/j.adaj.2019.09.011. PMID 31761029
- [Background] Al-Hadidi F, Bsisu I, AlRyalat SA, Al-Zu'bi B, Bsisu R, Hamdan M, Kanaan T, Yasin M, Samarah O. Association between mobile phone use and neck pain in university students: A cross-sectional study using numeric rating scale for evaluation of neck pain. PLoS One. 2019 May 20;14(5):e0217231. doi: 10.1371/journal.pone.0217231. eCollection 2019. PMID 31107910
- [Background] Mkontwana N, Novikova N. Oral analgesia for relieving post-caesarean pain. Cochrane Database Syst Rev. 2015 Mar 29;2015(3):CD010450. doi: 10.1002/14651858.CD010450.pub2. PMID 25821010